CLINICAL TRIAL: NCT04129619
Title: A Double-Blind, Placebo-Controlled, Phase 2, Responsive Adaptive Randomization Study of ORP-101 in Patients With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: A Comparison of the Effects of ORP-101 Versus Placebo in Adult Patients With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrphoMed, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: OM-201
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ORP-101 50 mg (Experimental): ORP-101 (50 mg) once daily
  Interventions: Drug: ORP-101
- ORP-101 100 mg (Experimental): ORP-101 (100 mg), once daily
  Interventions: Drug: ORP-101
- Placebo (Placebo Comparator): Matching placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORP-101 — Oral tablet
  Other Names: dibuprenorphine-ethyl-ether
  Arms: ORP-101 100 mg; ORP-101 50 mg
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of ORP-101 versus placebo on stool consistency and abdominal pain in patients with Irritable Bowel Syndrome with Diarrhea (IBS-D). It will also assess the safety and tolerability of ORP-101 in patients with IBS-D.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the efficacy, safety and tolerability of ORP-101 in patients with IBS-D. This is a randomized, double-blind, placebo-controlled, 3-arm, 12-week, parallel proof-of-concept study with 2 active arms (50 mg and 100 mg ORP-101, QD) and 1 matching placebo arm, using a responsive adaptive randomization approach. After screening, patients who qualify will enter the baseline symptom assessment period, during which they will be instructed on completion of an electronic diary for daily collection of data related to their IBS symptoms, bowel function and loperamide rescue usage (not allowed during baseline).

Patients who meet all entry criteria will be randomized to receive one of two different doses of ORP-101 tablets or placebo for 12 weeks. The study drug will be taken once daily, approximately 30 minutes prior to breakfast. Patients will return to the clinic on Days 14, 28, 56, 84 (12 weeks) and 2 weeks after dosing has completed (Day 98) for a follow-up visit.

Study subjects will include both male and female adults. Approximately 320 patients with IBS-D will be randomized to receive study drug or placebo. Randomization will be stratified by history of cholecystectomy/gallbladder agenesis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with protocol, including completion of electronic daily diary as required.
* Has a diagnosis of IBS-D (Irritable Bowel Syndrome with Diarrhea) and meets the Rome IV Criteria, by history, for both IBS and IBS-D.
* Has abdominal pain intensity score, and stool consistency as determined by protocol and assessed by Investigator for the week prior to randomization.
* Has not used loperamide within the 14 days prior to randomization.
* Is on a stable diet for the past 12 weeks and is not planning to change lifestyle and/or diet during study.

Exclusion Criteria:

* History of clinically relevant pancreatic conditions including pancreatitis, pancreas divisum, or Sphincter of Oddi (SO) dysfunction with pancreatic manifestations.
* History of biliary pathology including acute cholecystitis within 6 months or biliary pain including post-cholecystectomy pain.
* Patients who have had biliary sphincterotomy with post-procedure persistent abnormal liver function transaminases (LFTs).
* Planned elective surgery within the next 4 months.
* Significant and/or severe medical illnesses such as cardiovascular, neurological, infectious, renal, hepatic or respiratory disorders that would interfere with the patient's medical care, participation in, or conduct of the study.
* History of intestinal obstruction, stricture, toxic megacolon, GI (gastro-intestinal) perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (e.g. aorto-iliac disease).
* History of lactose intolerance uncontrolled on a lactose-free diet, or other malabsorption syndromes (e.g. fructose malabsorption).
* Dysphagia or difficulty swallowing pills.
* History of inflammatory bowel disease, celiac disease, Clostridium difficile colitis or have had recent unexplained GI bleeding within 3 months prior to screening.
* History of major gastric, hepatic, pancreatic or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy allowed as long as occurred > 3 months prior to trial screening; uncomplicated laparoscopic or open cholecystectomy is allowed if no history of post-operative biliary tract pain and surgery occurred > 3 months prior to screening).
* Patients >40 years of age at high risk for colon cancer must have had a screening colonoscopy within the past 3 years prior to trial screening visit or > 50 years of age, must have had a normal screening colonoscopy within the past 10 years prior to trial screening visit. Patients with Lynch Syndrome or Familial Polyposis are excluded from the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Are Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain and Daily Stool Consistency Scores | Week 12
  Composite responders are defined as participants who met the daily response criteria for at least 50% of the days with diary entries over the 12-week interval. A participant must meet both of the following criteria on a given day to be a daily responder: 1) Daily pain response: worst abdominal pain scores in the past 24 hours improved by ≥30% compared to baseline (average of daily worst abdominal pain the week prior to randomization). 2) Average of daily stool consistency response for all reported bowel movements on the specific day: Bristol Stool Scale (BSS) score <5 (ie, score of 1, 2, 3, or 4) or the absence of a bowel movement if accompanied by ≥30% improvement in worst abdominal pain compared to baseline pain.

SECONDARY OUTCOMES:
Percentage of Participants Who Are Responders in Daily Worst Abdominal Pain Scores | Week 12
  Pain responders over the interval from Weeks 1-12 are defined as those patients who meet the daily pain response criteria for at least 50% of days with diary entry during the interval. To be eligible to be a responder, a patient must have a minimum of 60 days of diary entries over the 12-week interval.
Percentage of Participants Who Are Responders in Daily Stool Consistency Scores | Baseline to Week 12
  Stool consistency responders over the interval from Weeks 1-12 are defined as those patients who meet the daily stool consistency response criteria for at least 50% of days with diary entry during the interval. To be eligible to be a responder, a patient must have a minimum of 60 days of diary entries over the 12-week interval.
Percentage of Participants Who are Responders in IBS Global Symptom Scores | Week 12
  IBS Global Symptom Score: Change from baseline for interval from Weeks 1-12: A responder is defined as a patient who has an IBS global symptom score of 0 (none) or 1 (mild) or daily IBS symptom score improved by ≥ 2.0 compared to the average in the week prior to randomization. A minimum of 60 days of diary entries over the 12-week interval is required for responders.
Percentage of Participants Who are Responders in IBS Adequate Relief Scores | Week 12
  IBS Adequate Relief: Percent of responders over the interval from Weeks 1-12. Responders are defined as those patients with a weekly response of "Yes" to adequate relief of their IBS symptoms for at least 50% of the total weeks during the interval.
Percentage of Participants Who Are Modified Composite Responders Based on Responder Endpoints | Week 12
  A modified composite responder endpoint in which a daily responder will be defined as having both: 1) Pain response: worst abdominal pain score in the past 24 hours improved ≥ 30% compared to the average in the week prior to randomization. 2) Stool consistency response: all bowel movements on the specific day must have BSFS score < 5 or the absence of a bowel movement if accompanied by ≥ 30% improvement in worst abdominal pain.
Change from Baseline in Daily Abdominal Discomfort Scores | Week 12
  Discomfort: Change from baseline in daily abdominal discomfort scores
Change from Baseline in Daily Abdominal Bloating Scores | Week 12
  Bloating: Change from baseline in daily abdominal bloating scores
Number of Bowel Movements Per Day | Week 12
  Frequency: Change from baseline in mean number of bowel movements per day
Number of Bowel Incontinence Free Days | Week 12
  Change from baseline in mean number of bowel incontinence episodes per day as well as the number of incontinence-free days

CONTACTS AND LOCATIONS:
Locations (74):
- United States (74):
  - Achieve Clinical Research (Site 155), Birmingham, Alabama
  - Synexus Clinical Research US, Inc. - Phoenix Southeast (Site 123), Chandler, Arizona
  - Elite Clinical Studies - Phoenix (Site 116), Phoenix, Arizona
  - Del Sol Research Management - BTC (Site 165), Tucson, Arizona
  - Synexus Clinical Research US, Inc. - Orange Grove Family Practice (Site 118), Tucson, Arizona
  - Del Sol Research Management - BTC (Site 130), Tucson, Arizona
  - Preferred Research Partners - ClinEdge (Site 103), Little Rock, Arkansas
  - Applied Research Center (Site 158), Little Rock, Arkansas
  - Connecticut Clinical Research Foundation (Site 136), Bristol, Connecticut
  - Imagine Research of Palm Beach County (Site 187), Boynton Beach, Florida
  - Meridien Research - Lakeland (Site 167), Lakeland, Florida
  - Precision Clinical Research LLC (Site 139), Lauderdale Lakes, Florida
  - Meridien Research, Maitland - Inpatient (Site 141), Maitland, Florida
  - Oviedo Medical Research (Site 140), Oviedo, Florida
  - Clinical Research Center of Florida (Site 186), Pompano Beach, Florida
  - Meridien Research - St. Petersburg (Site 132), St. Petersburg, Florida
  - Agile Clinical Research Trials, LLC (Site 163), Atlanta, Georgia
  - Gastrointestinal Diseases, Inc. Research (Site 137), Columbus, Georgia
  - Meridian Clinical Research (Site 169), Savannah, Georgia
  - In Quest Medical Research, LLC (Site 131), Suwanee, Georgia
  - GNP Research (Site 145), Valdosta, Georgia
  - Northwest Clinical Trials - ClinEdge (Site 133), Boise, Idaho
  - Synexus Clinical Research US, Inc. - Chicago (Site 120), Chicago, Illinois
  - Investigators Research Group, LLC (Site 188), Brownsburg, Indiana
  - Synexus Clinical Research US, Inc. - Allaw (Site 102), Evansville, Indiana
  - Alliance for Multispecialty Research, LLC (Site 159), Wichita, Kansas
  - Beth Israel Deaconess Medical Center (Site 115), Boston, Massachusetts
  - AES-DRS-Synexus Clinical Research US, Inc.-Minneapolis (site 114), Richfield, Minnesota
  - Sundance Clinical Research (Site 175), St Louis, Missouri
  - Synexus Clinical Research US, Inc. - Omaha (Site 113), Omaha, Nebraska
  - Synexus Clinical Research US, Inc. - McGill Family Practice, P.C. (Site 126), Papillion, Nebraska
  - Jubilee Clinical Research - BTC (Site 162), Las Vegas, Nevada
  - Sierra Clinical Research (Site 179), Las Vegas, Nevada
  - Lovelace Scientific Resources Inc. (Site 176), Albuquerque, New Mexico
  - NY Scientific (Site 153), Brooklyn, New York
  - Long Island Gastrointestinal Research Group LLP (Site 107), Great Neck, New York
  - Synexus Clinical Research US, Inc. - Queens (Site 119), Jamaica, New York
  - Mid Hudson Medical Research PLLC (Site 174), Newburgh, New York
  - Upstate Clinical Research Associates LLC - ClinEdge (Site 164), Williamsville, New York
  - OnSite Clinical Solutions, LLC - ClinEdge (Site 147), Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC - ClinEdge (Site 146), Charlotte, North Carolina
  - Peters Medical Research, LLC - ClinEdge (SIte 111), High Point, North Carolina
  - PMG Research of Salisbury LLC (Site 110), Salisbury, North Carolina
  - PMG Research of Wilmington (Site 185), Wilmington, North Carolina
  - PMG Research of Winston-Salem (Site 124), Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc. - Akron (Site 122), Akron, Ohio
  - Hometown Urgent Care and Research (Site 150), Cincinnati, Ohio
  - Synexus Clinical Research US, Inc. - Cincinnati (Site 127), Cincinnati, Ohio
  - Synexus Clinical Research US, Inc. - Columbus (Site 108), Columbus, Ohio
  - Hometown Urgent Care and Research (Site 149), Columbus, Ohio
  - Remington Davis Inc (Site 144), Columbus, Ohio
  - PriMed Clinical Research - ClinEdge (Site 121), Dayton, Ohio
  - Hometown Urgent Care and Research (Site 151), Dayton, Ohio
  - Medical Research international (Site 180), Oklahoma City, Oklahoma
  - Tristar Clinical Investigations, P.C. (Site 168), Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC (Site 171), Uniontown, Pennsylvania
  - Piedmont Research Partners LLC - BTC (Site 157), Fort Mill, South Carolina
  - Synexus clinical Research US, Inc. - Greer (Site 105), Greer, South Carolina
  - WR-ClinSearch, LLC (Site 129), Chattanooga, Tennessee
  - The Jackson Clinic PA - ClinEdge (Site 135), Jackson, Tennessee
  - New Phase Research & Development (Site 181), Knoxville, Tennessee
  - Benchmark Research - Austin (Site 178), Austin, Texas
  - Advanced Medical Trials (SIte 142), Georgetown, Texas
  - Pioneer Research Solutions (Site 125), Houston, Texas
  - Synergy Group US, LLC - Missouri City - Hunt (Site 156), Missouri City, Texas
  - DM Clinical Research - LinQ Research - ERN (Site 109), Pearland, Texas
  - Synexus Clinical Research US, Inc. - San Antonio (Site 112), San Antonio, Texas
  - Clinical Trials of Texas Incorporated - ClinEdge (Site 134), San Antonio, Texas
  - Synexus Clinical Research US, Inc. - Salt Lake City (Site 101), Murray, Utah
  - Advanced Research Institute (Site 117), Ogden, Utah
  - Health Research of Hampton Roads Inc. (Site 173), Newport News, Virginia
  - The Center of Gastrointestinal Health (Site 152), Petersburg, Virginia
  - Northwest Clinical Research Center - ClinEdge (Site 148), Bellevue, Washington
  - Exemplar Research, Inc. - Morgantown (Site 172), Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm